CLINICAL TRIAL: NCT05893680
Title: Comparison of the Effects of Online Games, Cold Applications and Placebo in Reducing Pain in Children Undergoing Orthopedic and Traumatology Surgery
Brief Title: Nonpharmacological Management of Postoperative Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İlke Karabıyık (Other)
Responsible Party: Sponsor-Investigator, İlke Karabıyık, Nurse, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1122
Record Dates: First submitted 2023-04-08; First posted 2023-06-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Orthopedic Disorder; Post Operative Pain
Keywords: postoperative pain; orthopedic and traumatology surgery; pediatri; cold application; placebo; online games
MeSH Terms: conditions — Musculoskeletal Diseases; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled experiment to compare the effects of cold application, online gaming, and placebo on postoperative pain in children. Participants who met the selection criteria were randomly assigned to the "online gaming," "cold application," "placebo," and "online gaming and cold application" groups through a pre-determined lottery. Subsequently, the pain-reducing intervention specific to the assigned group was applied to the child who was randomized to that group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group to play online games (Experimental): The child's pain was evaluated 4 hours after the surgery, and then he/she was allowed to play an online game that he/she knew, loved, and wanted to play for 20 minutes.
  Interventions: Other: Group to play online games
- Group that received cold application (Experimental): The child's pain was evaluated 4 hours after the surgery, and then a clean gauze wrapped cold gel pack was applied to the surgical site for 20 minutes.
  Interventions: Other: Group that received cold application
- Group that received placebo (Placebo Comparator): The child in the relevant group had their pain evaluated 4 hours after the surgery, and then was given 2 cc of 0.9% saline (isotonic) solution intravenously, while being told that it was a painkiller administered to both the child and the parent.
  Interventions: Drug: Group that received placebo (PHYSIOLOGICAL SALINE ISOTONIC 9 mg/ml AMPULE)
- "Group that played an online game and received cold application at the same time (Active Comparator): Pain assessment was performed on the child in the relevant group 4 hours after surgery, and then while playing an online game that the child knew, liked, and wanted to play, a clean gauze-wrapped cold gel pack was applied to the surgical site for cold therapy. The interventions lasted for 20 minutes.
  Interventions: Other: Group that played an online game and received cold application at the same time

INTERVENTIONS:
Other: Group to play online games — Playing games in children is one of the non-pharmacological pain relief methods. In this study, the effect of playing an online game on pain level in children who underwent orthopedic surgery for pain management after the surgery was measured.
  Arms: Group to play online games
Other: Group that received cold application — Previous studies have demonstrated that cold application has anti-inflammatory, muscle spasm reducing, and pain relieving properties. In this study, the effect of cold application on pain level in children who underwent orthopedic surgery was investigated.
  Arms: Group that received cold application
Drug: Group that received placebo (PHYSIOLOGICAL SALINE ISOTONIC 9 mg/ml AMPULE) — The placebo effect has been demonstrated in various studies today. Some of these studies describe placebo analgesia. In this study, the placebo analgesic effect was investigated, and the child and parent were told that an analgesic was applied, but instead 2 cc of PF 0.9% ISOTONIC SODIUM CHLORIDE solution was intravenously administered.
  Other Names: PHYSIOLOGICAL SALINE ISOTONIC 9 mg/ml AMPULE
  Arms: Group that received placebo
Other: Group that played an online game and received cold application at the same time — To investigate the combined effect of online gaming and cold application as two separate non-pharmacological interventions, both interventions were applied together in this group
  Arms: "Group that played an online game and received cold application at the same time

SUMMARY:
The 3 non-pharmacological methods of online gaming, cold application, and placebo were chosen to reduce postoperative pain in children undergoing orthopedic and traumatology surgery. The effect of these 3 non-pharmacological methods on pain reduction was measured and compared.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial to compare the effects of cold application, online gaming, and placebo on postoperative pain in children.

The sample size of the study was determined as 160 children, considering a 5% alpha error rate, 90% power, and the probability of loss of data during data collection, using G*Power program (3.1.9.2.) According to this result, the population of the study is planned to be formed with 160 child patients, aged between 7-12, who are hospitalized in the Palace Lower Floor Orthopedics Service of Istanbul Metin Sabancı Baltalimanı Bone Diseases Training and Research Hospital. The 160 children who make up the sample will be randomly assigned to "online game and cold application", "online game", "cold application", and "placebo" groups, previously sorted as group 1, group 2, group 3, and group 4 by the lottery method. In the study, the intervention of the relevant group will be applied to each child during pain control in each group.

A randomization list consisting of 40 blocks of four, based on age, gender, and the extremity region where the operation was performed, was created (https://www.randomizer.org/#randomize) to assign the children participating in the study to the groups randomly.

After the children were assigned to the intervention groups homogeneously and randomly, the study was started.

Before applying any pain-reducing interventions to all children in all the intervention groups, pain assessment was conducted using the visual analog scale (VAS) at 4 hours after surgery. The child's parent was also asked to evaluate the child's pain independently using the same scale. In this way, pre-intervention pain assessment was performed. Later, the pain-reducing intervention specific to the group in which the child was randomized was applied to the child.

The cold application group received a 20-minute application of cold gel that had been kept in the freezer for at least 2 hours on the surgical site of the children.

The children in the online game group were allowed to play a game they knew and wanted to play beforehand. This intervention lasted for 20 minutes.

The children in the group receiving both cold application and online game intervention were provided with the opportunity to play a previously known and desired online game while applying cold gel that had been kept in the freezer for at least 2 hours to the surgical site for 20 minutes. The intervention lasted for 20 minutes.

The children in the placebo group were administered 2 ml dose of sterile %0.9 saline solution (isotonic) intravenously. The mother and child were informed that the intervention administered during the procedure was a pain reliever.

After starting the pain-reducing interventions in all groups, pain assessment using VAS was repeated at 10 and 20 minutes with a double-blind technique by asking both the child and the parent. The cold application and online game interventions were stopped after the pain assessment at 20 minutes. Then, pain measurement with VAS was repeated at 40 minutes after the start of the pain-reducing interventions, and the measurement results were recorded to end the study.

In all groups, routine monitoring of fever, pulse, respiration, and saturation, which are already part of the clinic's standard practice, has been performed.

The assumptions of parametric tests for the obtained data will be evaluated to determine the appropriate statistical method, and data analysis will be performed. The results of the analysis will be interpreted, and the relevant data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 7-12 age group
* Having undergone lower or upper extremity surgery
* Receiving general anesthesia during surgery
* Having a body temperature not higher than 37.5°C
* Those who are hospitalized in the orthopedic service and agree to participate along with their parents.

Exclusion Criteria:

* After the surgery, children who had intense pain in the first 4 hours and were given analgesics, children under 7 or over 12 years old, children with a fracture in the active arm for the online game group, children with a fever above 37.5°C, patients who were not fully recovered at 4 hours after the surgery and could not communicate, patients with mental motor development retardation, patients with plaster treatment for the cold application group, patients who received botulinum toxin injection during surgery and patients who underwent biopsy will be excluded from the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Statistical analysis | 8 months
  The data will be analyzed by deciding on the relevant statistical method by evaluating whether the assumptions of parametric tests are met. The analysis results will be interpreted, and the relevant data will be recorded.

SECONDARY OUTCOMES:
Body weight | 8 months
  Body weight" refers to the measure of a person's or animal's mass or weight. The measurement was made with a scale in kilograms.
Height | 8 months
  Height refers to the vertical measurement of a person, typically measured from the bottom of the feet to the top of the head, usually expressed in units of centimeters (cm) or feet and inches (ft/in). It is commonly used as an indicator of physical growth and development. The height was measured with a measuring tool and recorded in cm.
pulse | 8 months
  Pulse, refers to the rhythmic expansion and contraction of the arteries as blood is pumped through the body by the heart. It can be felt as a beat in different parts of the body, such as the wrist, neck, or ankle, and is typically measured in beats per minute (bpm). Pulse rate is an important clinical indicator of heart health and can be affected by various factors, including exercise, stress, and illness.
respiration | 8 months
  Respiration refers to the process of inhaling and exhaling air in and out of the lungs, which facilitates the exchange of oxygen and carbon dioxide in the body.
body temperature | 8 months
  Body temperature refers to the average temperature of the body, typically measured in degrees Celsius (°C) or Fahrenheit (°F). It is an important indicator of overall health and can be measured in various ways, such as with a thermometer. Normal body temperature typically ranges from 36.5°C to 37.5°C (97.7°F to 99.5°F). In this study, body temperature was measured using a thermometer and recorded in degrees Celsius.
saturation | 8 months
  Saturation refers to the level or amount of a particular substance or component in a mixture or solution. It can also refer to the degree of oxygen saturation in the blood, which is a measure of the percentage of hemoglobin molecules carrying oxygen in the blood. The values were recorded by measuring with a pulse oximeter.

OTHER OUTCOMES:
pain assessment | 8 months
  Pain assessment refers to the process of evaluating the severity and characteristics of a person's pain. It involves assessing the location, intensity, duration, and other factors that contribute to the pain experience. Pain assessment helps healthcare professionals determine the most appropriate pain management strategies for a patient. In this study, visual analog scale was used. The VAS (Visual Analog Scale) consists of a straight line measuring 100 mm. The endpoints of the line are labeled as 0 (no pain at all) and 10 (worst imaginable pain). With this scale, the child is asked to mark a point between 0 and 10 or verbally express the level of their pain to assess pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: İlke Karabıyık, Principal Investigator — İstanbulUC
Locations (1):
- Istanbul Metin Sabancı Baltalimanı Bone Diseases Training and Research Hospital., Istanbul, Istanbul/Sarıyer, Turkey (Türkiye)